CLINICAL TRIAL: NCT02116023
Title: The Effect of Different Doses of Processed Whole Orange on Subjective Ratings of Satiety
Brief Title: The Effects of Processed Whole Orange on Subjective Ratings of Satiety
Acronym: POAS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PepsiCo Global R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: PEP-1402
Record Dates: First submitted 2014-04-10; First posted 2014-04-16 (Estimated); Last update posted 2014-10-28 (Estimated); Status verified 2014-10

CONDITIONS: Self Reported Ratings of Hunger
Keywords: Satiety, beverage, crossover

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Orange flavored beverage - Test1 (Experimental): 240ml processed whole orange low dose
  Interventions: Other: Orange flavored beverage
- Orange flavored beverage - Test2 (Experimental): 240ml processed whole orange high dose
  Interventions: Other: Orange flavored beverage
- Orange flavored beverage - Placebo (Placebo Comparator): 240ml orange beverage
  Interventions: Other: Orange flavored beverage

INTERVENTIONS:
Other: Orange flavored beverage

SUMMARY:
The study is a human dietary test meal study that is a randomized, controlled, double blind, cross over design with 3 intervention arms that will investigate the subjective ratings of satiety in response to different levels of processed whole orange compared with a sugar-matched isocaloric control

ELIGIBILITY:
Inclusion Criteria:

* Gender: male or female
* Age at start of the study: males and females ≥ 21and ≤ 65 years
* Females taking contraceptive pill or post menopausal
* Body Mass Index (BMI) ≥ 18.5 and ≤ 27 kg/m2
* Apparently healthy: measured by questionnaire, no reported current or previous -metabolic diseases or chronic gastrointestinal disorders
* Reported dietary habits: no medically prescribed diet, no slimming diet within the past 3 months, used to eating 3 meals a day
* Reported intense sporting activities ≤ 10h/w
* Reported alcohol consumption ≤21 units/w Informed consent signed
* Recruitment form filled out

Exclusion Criteria:

* Smoking
* Premenopausal females not taking the contraceptive pill
* Dislike, allergy or intolerance to test products
* Possible eating disorder (measured by SCOFF questionnaire score >1)
* Eating habits questionnaire score >14
* Reported medical treatment that may affect eating habits/satiety
* Food allergies or intolerance

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-03; Primary Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Self reported ratings of hunger and fullness | 0-2 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, United Kingdom